CLINICAL TRIAL: NCT01809587
Title: Open Label Study to Assess the Safety and Efficacy of IQP-PO-101 in Regulating Bowel Movement Frequency
Brief Title: IQP-PO-101 for the Regulation of Bowel Movement Frequency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INQ/026612
Record Dates: First submitted 2013-03-07; First posted 2013-03-12 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Constipation; Irregular Bowel Movement Frequency
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IQP-PO-101 (Experimental): Day 1 to Day 7 - 1 sachet to be mixed in 250ml of water and consumed twice a day Day 8 to Day 28 - 1 sachet to be mixed in 250ml of water and consumed once a day Day 28 to Day 42 - no investigational product intake (post treatment observation only)
  Interventions: Device: IQP-PO-101

INTERVENTIONS:
Device: IQP-PO-101

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of IQP-PO-101 in regulating the bowel movement frequency

ELIGIBILITY:
Inclusion Criteria:

* A subject must have experienced 2 - 4 bowel movements per week and at least 2 of the following symptoms over the preceding 3 months (self-reported):

  * Excessive straining
  * Lumpy or hard stools
  * Sensation of anorectal obstruc-tion
  * A sense of incomplete evacua-tion of bowel movements
  * A need for digital manipulation to facilitate evacuation
* Recorded between 4 and 9 defecations in the 14-day bowel movement diary during the run-in period
* Subjects of childbearing potential must agree to use appropriate contraceptive methods during run-in and treatment period
* Commitment to avoid the use of any laxatives and/ or other medicinal products/ supplements that may interfere with bowel movement frequency during the run-in and treatment period
* Written informed consent.

Exclusion Criteria:

* Known sensitivity to the ingredients of the device
* Any organic gastrointestinal diseases, congenital or otherwise
* Presence of occult blood on screening
* Constipation that may have been drug-induced
* Use of any laxative/ products that help ease bowel movements within 7 days of the screening visit
* Constipation other than idiopathic constipation
* Presence of other factor(s) that, in the in-vestigator's judgement, should preclude subject participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Bowel movement frequency | 6 weeks
  Subjects will keep a record of the number of bowel movements, if any, from 00:00 hours to 23:59 hours (midnight to midnight) daily.

SECONDARY OUTCOMES:
Bristol Stool Form Scale | 6 weeks
  Subjects will keep a record of their stool form, for each bowel movement.
Straining at the start/ end of defecation | 6 weeks
  On a 100mm visual analogue scale (VAS), subjects will rate their feeling of straining at the start/ end of defecation for each bowel movement.
Pain during defecation | 6 weeks
  On a 100mm visual analogue scale (VAS), subjects will rate their pain during defeca-tion for each bowel movement.
Feeling of incomplete evacuation | 6 weeks
  With each bowel movement, subjects will mark "Yes" or "No" to indicate whether there was a feeling of incomplete evacuation.
Evaluation of efficacy by subjects | 4 weeks
  The subjects evaluate independently the efficacy of the investigational device (global scaled evaluation with "very good", "good", "moderate" and "poor").
Evaluation of efficacy by investigator | 4 weeks
  The investigator evaluates independently the efficacy of the investigational device (global scaled evaluation with "very good", "good", "moderate" and "poor")
Full blood count | 4 weeks
  Venous blood samples are obtained at screening and the end of the treatment period (4 weeks)
Clinical chemistry | 4 weeks
  Venous blood samples are obtained at screening and the end of the treatment period (4 weeks) for measurements of uric acid, HbA1c and lipid profiles. An analysis will be done based on the change between the 2 periods.
Safety evaluation by subjects | 4 weeks
  The subjects evaluate independently the safety of the investigational device (global scaled evaluation with "very good", "good", "moderate" and "poor")
Safety evaluation by investigators | 4 weeks
  The investigators evaluate independently the safety of the investigational device (global scaled evaluation with "very good", "good", "moderate" and "poor")
Adverse events | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Analyze & Realize Ag, Berlin, State of Berlin, Germany